CLINICAL TRIAL: NCT00663910
Title: Evaluation of Protoporphyrin Formation in Non-Melanoma Skin Cancers After Topical Application of 5-Aminolevulinic Acid: A Pilot Study
Brief Title: Topical Aminolevulinic Acid in Patients With Nonmelanoma Skin Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Of the 8 histologically proven tumors, detection of PpIX proved to be ambiguous.
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE-9Z07-CC417; P30CA043703 (NIH); P01CA084203 (NIH); CC417 (Other: Case Comprehensive Cancer IRB)
Record Dates: First submitted 2008-04-19; First posted 2008-04-22 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Non-melanomatous Skin Cancer
Keywords: basal cell carcinoma of the skin; squamous cell carcinoma of the skin; recurrent skin cancer
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms | interventions — Aminolevulinic Acid; Biopsy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Aminolevulinic Acid — On Day 1, ALA will then be applied topically to the center of the tumor surface (at the location of its greatest diameter) in a standardized manner with great care not to include normal skin. The solution will be applied directly to the lesions by dabbing gently with a wet applicator tip. Enough solution will be applied to uniformly wet the exposed lesion surface. Once the initial application has dried, the ALA will be applied again in the same manner. The ALA will be left on for 2 hours under occlusion with Duoderm Extra Thin®.
  Other Names: ALA
Procedure: biopsy — Then local anesthesia, lidocaine 1% with epinephrine 1:100,000, will be administered and before the tumor is excised by one of the Cleveland Clinic MOHS surgeons, a 2mm punch biopsy will be taken from the area where the ALA was previously applied. The punch biopsy will be full thickness, extending to the subcutaneous fat.
Procedure: diagnostic imaging technique — Two hours after the amniolevlulenic acid was applied, the measurements of surface fluorescence will be repeated with the hand held dosimeter.
  Other Names: Aurora dosimeter
Procedure: therapeutic conventional surgery — The non-melanoma skin cancer will be excised using the MOHS procedure.

SUMMARY:
RATIONALE: Studying samples of tumor tissue in the laboratory from patients with nonmelanoma skin cancer that has been treated with topical aminolevulinic acid may help doctors predict how patients will respond to photodynamic therapy.

PURPOSE: This clinical trial is studying topical aminolevulinic acid in patients with nonmelanoma skin cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the distribution and depth of protoporphyrin IX (PpIX) within different types of nonmelanoma skin cancers after topical aminolevulinic acid (ALA) administration.
* To obtain in vivo measurements of ALA-induced PpIX formation within different zones of the tumors as measured by fluorescence detection methods.
* To correlate the level of PpIX fluorescence detected by non-invasive optical measurements with morphological characteristics of the tumors.
* To establish a skin cancer tissue bank.

OUTLINE: Topical aminolevulinic acid (ALA) is applied to the center of the tumor surface. Patients then undergo punch tumor biopsy of the area where the ALA is applied followed by surgery to remove the tumor. Tissue samples are assessed for protoporphyrin (PpIX) levels by fluorescence confocal microscopy and hyperspectral imaging. Excess tumor tissue may be stored in a skin cancer tissue bank. Surface measurements (from a total of 5 surface sites) of PpIX fluorescence are taken at baseline and at 2 hours after ALA application using an optical fiber-based hand-held dosimeter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must have at least 1 biopsy-proven nonmelanoma skin cancer with a minimum diameter of 4 mm
* No tumors located on the eyelids, distal nose, cartilaginous portions of the ears, or lips

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known hypersensitivity to aminolevulinic acid or any component of this medication

PRIOR CONCURRENT THERAPY:

* Concurrent immunosuppressive or chemotherapeutic medications allowed
* Concurrent corticosteroids (taken by mouth or large doses taken with an inhaler) allowed
* Concurrent systemic retinoids (e.g., isotretinoin, acitretin, bexarotene, alitretinoin) or vitamin A allowed
* Other concurrent medications that may affect epidermal growth and differentiation (e.g., anti-EGFR monoclonal antibodies) allowed
* No concurrent participation in another clinical trial
* No concurrent topical treatment for the target tumor or for other nonmelanoma skin cancers
* No concurrent medical therapy or radiotherapy for other cancers

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Maximum depth of protoporphyrin IX (PpIX) fluorescence within different types of nonmelanoma skin cancers after topical aminolevulinic acid (ALA) administration | Day 1

SECONDARY OUTCOMES:
In vivo measurements of ALA-induced PpIX formation within different zones of the tumors as measured by fluorescence detection methods | Day 1
Correlation of the level of PpIX fluorescence detected by non-invasive optical measurements with morphological characteristics of the tumors | Day 1
Establishment of a skin cancer tissue bank | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Edward V. Maytin, MD, PhD, Study Chair — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.